CLINICAL TRIAL: NCT07328841
Title: Reduced-Dose Versus Conventional-Dose Intensity-Modulated Radiation Therapy in Locally Advanced Nasopharyngeal Carcinoma With Remission After Induction Chemotherapy and Immunotherapy: A Multicenter, Phase III Clinical Trial
Brief Title: Reduced-dose Versus Conventional-dose Intensity-modulated Radiation Therapy for Locally Advanced Nasopharyngeal Carcinoma With Remission After Induction Chemotherapy and Immunotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ming-Yuan Chen (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Professior, Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.BYAFZZX.043
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: Nasopharyngeal Carcinoma; Locally Advanced; Epstein-Barr Virus DNA; EBV DNA clearance; undetectable EBV DNA; reduced-dose radiotherapy; Randomized non-inferiority trial; Concurrent chemoradiotherapy; complete response; partial response; PD-1inhibitor
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Pathologic Complete Response | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction chemotherapy plus reduced-dose radiotherapy and concurrent chemotherapy (Experimental)
  Interventions: Drug: Full course of PD-1blockades; Drug: Cisplatin-based induction chemotherapy; Radiation: Reduced-dose radiotherapy; Drug: Concurrent Chemotherapy
- Induction chemotherapy plus conventional concurrent chemoradiotherapy (Active Comparator)
  Interventions: Drug: Full course of PD-1blockades; Drug: Cisplatin-based induction chemotherapy; Radiation: Standard-dose radiotherapy; Drug: Concurrent Chemotherapy

INTERVENTIONS:
Drug: Full course of PD-1blockades — Toripalimab 240 mg, once every 3 weeks (Q3W), intravenous infusion (iv). A total of 12 courses of treatment will be administered, including 3 courses during the induction chemotherapy phase, 3 courses during the radiotherapy phase, and 6 courses during the post-radiotherapy maintenance phase. Administration will start on Day 1 of induction chemotherapy and continue after the end of radiotherapy until the occurrence of intolerable toxicities, disease progression, withdrawal of consent, determination by the investigator that the patient needs to withdraw from treatment, or the completion of 12 courses, whichever comes first.
Drug: Cisplatin-based induction chemotherapy — Cisplatin-based induction chemotherapy will be given every 3 weeks for 3 cycles before radiotherapy.
Radiation: Standard-dose radiotherapy — GTVnx/nd:69.96Gy/33Fr/2.12Gy CTV1: 59.4Gy/33Fr/1.8Gy CTV2: 54.12Gy/33Fr/1.64Gy
  Arms: Induction chemotherapy plus conventional concurrent chemoradiotherapy
Radiation: Reduced-dose radiotherapy — GTVnx/nd:63.6Gy/30Fr/2.12Gy CTV1: 54Gy/30Fr/1.8Gy CTV2: 49.2Gy/30Fr/1.64Gy
  Arms: Induction chemotherapy plus reduced-dose radiotherapy and concurrent chemotherapy
Drug: Concurrent Chemotherapy — Cisplatin 100mg/m2 every 3 weeks for 2 cycles

SUMMARY:
To explore the efficacy and safety of reduced-dose radiotherapy combined with concurrent chemotherapy and immunotherapy in stage Ⅳa (AJCC 8th,) locally advanced nasopharyngeal carcinoma patients who are sensitive to induction chemoimmunotherapy (assessed as complete response [CR]/partial response [PR] by imaging, with EBV DNA copy number reduced to zero or below the lower limit of detection), so as to provide a new treatment option for these patients.

DETAILED DESCRIPTION:
In a prospective clinical trial, under full-course immunotherapy, a platinum-based chemotherapy combined with immunotherapy regimen is used as the induction treatment protocol. Patients with stage Ⅳa (AJCC 8th,) nasopharyngeal carcinoma who achieve partial response (PR) or complete response (CR) after induction treatment, with EBV DNA reduced to zero or below the lower limit of detection, are randomized at a 1:1 ratio. One group receives reduced-dose radiotherapy combined with concurrent chemoimmunotherapy, while the other group receives conventional-dose radiotherapy combined with concurrent chemoimmunotherapy.

Through follow-up, the differences in survival prognosis, incidence of complications, and quality of life between the two groups are observed. The aim is to evaluate whether, on the premise of ensuring non-inferior 3-year progression-free survival (PFS), reduced-dose radiotherapy shows superiority or significant improvement in ≥ grade 3 radiotherapy-related toxicities (especially xerostomia, dysphagia, and hearing loss) and quality of life. Thereby, it explores whether the treatment strategy of further reduced-dose radiotherapy is suitable for patients with locally advanced nasopharyngeal carcinoma who achieve CR/PR on imaging evaluation and have EBV DNA reduced to zero after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed nasopharyngeal non-keratinizing carcinoma (differentiated or undifferentiated type, i.e., WHO classification Type II or Type III).
2. Clinical stage: AJCC 8th edition staging: T4N0-2M0, T1-4N3M0 (stage IVa); AJCC 9th edition staging: T4N0-2M0, T1-4N3M0 (stage III).
3. After 3 courses of platinum-based chemotherapy combined with immunotherapy as induction treatment, the efficacy is assessed as PR or CR by nasopharyngoscopy and enhanced MRI of nasopharynx + neck, with EBV DNA reduced to zero or below the lower limit of detection.
4. Age: 18-70 years old.
5. PS/ECOG score (performance status score of 0 or 1).
6. Adequate organ function:

   1. Hematology: White blood cell count ≥ 4000/μL, neutrophil count ≥ 2000/μL, hemoglobin ≥ 9 g/dL, platelet count ≥ 100000/μL;
   2. Liver function: Bilirubin ≤ 1.5 × upper limit of normal (ULN) (patients with known Gilbert's disease and serum bilirubin level ≤ 3 × ULN are eligible), AST and ALT ≤ 1.5 × ULN, and alkaline phosphatase ≤ 1.5 × ULN; albumin ≥ 3 g/dL;
   3. Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min calculated by the Cockcroft-Gault formula.
   4. Proteinuria: Urine protein/creatinine ratio (UPC ratio) < 1.0. For those with UPC ratio ≤ 0.5, no further examination is required; for those with UPC ratio > 0.5, further testing showing 24-hour urine protein < 1000 mg is eligible.

   Note: The UPC ratio of random urine is an estimate of 24-hour urine protein quantification, and the two have a good correlation. The UPC ratio can be calculated using the following formulas:

   i. Urine protein/urine creatinine (if both protein and creatinine are in mg/dL); ii. (Urine protein) × 0.088/urine creatinine (if urine creatinine is in mmol/L).

   e) Coagulation function: International normalized ratio (INR) ≤ 1.5, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
7. Patients have signed the informed consent form and are willing and able to comply with the study's scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Patients whose laboratory test results within 7 days before enrollment do not meet the relevant standards.
2. Patients with efficacy evaluation of stable disease (SD) or progressive disease (PD) after 3 courses of platinum-based chemotherapy combined with immunotherapy as induction treatment, or whose EBV DNA has not been reduced to zero or below the lower limit of detection.
3. Patients who have received any of the following for primary lesions and/or cervical metastatic lesions: chemotherapy, immunotherapy, targeted therapy, or surgical treatment (excluding diagnostic treatment).
4. Patients with tumors accompanied by obvious liquefaction necrosis, which are unsuitable for radiotherapy or may lead to radioresistance.
5. Patients with tumors invading the brain parenchyma.
6. Patients with a history of severe allergic reactions to any components of other monoclonal antibodies or PD-1/PD-L1 monoclonal antibodies.
7. Patients with known or suspected autoimmune diseases, including dementia and epileptic seizures.
8. Patients with recurrence, distant metastasis, or concurrent other malignant tumors.
9. Patients with severe heart disease, pulmonary dysfunction, or cardiac/pulmonary function grade 3 or lower (including grade 3).
10. Patients with previous use of anti-PD-1/PD-L1 antibodies, anti-CTLA-4 antibodies, or any other antibodies acting on T-cell costimulatory or checkpoint pathways.
11. Patients with comorbidities requiring long-term treatment with immunosuppressive drugs or systemic/local use of corticosteroids at immunosuppressive doses before enrollment.
12. Patients with HIV positivity; HBsAg positivity with positive HBV DNA copy number (quantitative detection ≥ 1000 cps/ml); positive screening for chronic hepatitis C (HCV antibody positivity).
13. Patients with a history of allergic reactions to the drugs used in this study (gemcitabine, docetaxel, taxanes, cisplatin).
14. Patients with active tuberculosis (TB) who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening.
15. Patients who, within 4 weeks before enrollment: have received systemic or local glucocorticoid treatment, been vaccinated with any anti-infective vaccines (such as influenza vaccine, varicella vaccine, etc.), or used traditional Chinese herbal medicines with anti-tumor effects.
16. Women of childbearing age with positive pregnancy test results and lactating women.
17. Other patients deemed unsuitable for inclusion by the attending physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Progress-Free Survival (PFS) | 3 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Defined as the time interval from randomization to death due to any cause.
Locoregional Relapse-Free Survival (LRRFS) | 3 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Distant Metastasis-Free Survival (DMFS) | 3 years
  Defined as the time interval from randomisation to the date of first distant metastases.
Objective Response Rate (ORR) | assessed at 3 months after the end of concurrent chemoradiotherapy
  Defined as the proportion of patients with tumor reduction achieving complete response (CR) or partial response (PR), assessed at 3 months after the end of concurrent chemoradiotherapy.
The proportion of patients with treatment related acute complications | 1 year
  The proportion of patients with treatment related acute complications according to NCI-CTC5.0 criteria and RTOG criteria.
The proportion of patients with treatment related late complications | 3 years
  The proportion of patients with treatment related late complications according to NCI-CTC5.0 criteria and RTOG criteria.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (12):
- China (12):
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University cancer center, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Sun Yat-sen University (SYSU), Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Central South University Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Guangdong, Zhuhai